CLINICAL TRIAL: NCT04231955
Title: Comparison of Different Pain Rating Scales in Patients With Symptomatif Teeth
Brief Title: Comparison of Different Pain Rating Scales in Patients With Symptomatic Teeth
Acronym: CoPRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Tan Firat Eyuboglu, Assistant professor, Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 338
Record Dates: First submitted 2019-12-09; First posted 2020-01-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Pain; Dental Pain
Keywords: numerical rating scale; visual analogue scale; color analogue scale; faces rating scale; pain intensity
MeSH Terms: conditions — Pain; Toothache

STUDY DESIGN:
Intervention Model Description: all 50 patients marked their pain intensity levels of their relevant tooth in four different rating scales.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pain rating scales (Experimental): patients were asked to marked their pain intensity level on numerical rating scale between 0 and 10, on visual analogue scale, a straight line with one end indicating "no pain" and the other end indicating "worst pain possible". on color analogue scale, a straight line with one end indicating "no pain" and the other end indicating "worst pain possible"and color change towards to "worst pain possible" end and on a faces rating scale which consisted of six different faces representing different levels of pain intensity with the first face indicating "no pain" whilst last face indicating "worst pain possible". The result was recorded as pain intensity level.
  Interventions: Diagnostic Test: numerical rating scale; Other: visual analogue scale; Other: color analogue scale; Other: faces rating scale

INTERVENTIONS:
Diagnostic Test: numerical rating scale — patients were asked to marked their pain intensity level on numerical rating scale between 0 and 10 and the result was recorded as pain intensity level.
  Other Names: NRS
Other: visual analogue scale — Patients were asked to marked their pain intensity level on visual analogue scale, a straight line with one end indicating "no pain" and the other end indicating "worst pain possible". Then the distance between no pain end and patients' mark was measured and recorded as pain intensity level.
  Other Names: VAS
Other: color analogue scale — Patients were asked to marked their pain intensity level on color analogue scale, a straight line with one end indicating "no pain" and the other end indicating "worst pain possible"and color change towards to "worst pain possible" end. Then the distance between no pain end and patients' mark was measured and recorded as pain intensity level.
  Other Names: CAS
Other: faces rating scale — Patients were asked marked their pain on a faces rating scale which consisted of six different faces representing different levels of pain intensity with the first face indicating "no pain" whilst last face indicating "worst pain possible". The result was recorded as pain intensity level.
  Other Names: FRS

SUMMARY:
Patients with symptomatic teeth who applied endodontic clinic between April 2019 and December 2019 for root canal treatment were enrolled in this study. All patients were asked to fill four different rating scales: numerical rating scale, visual analogue scale, color analogue scale and faces rating scale for their relevant tooth which is symptomatic and need of root canal treatment. The four scales were then compared statistically.

DETAILED DESCRIPTION:
50 patients who applied endodontic clinic between April 2019 and December 2019 and had symptomatic teeth which were in need of root canal treatment were enrolled for this study. Study detail were explained to all patients and they were then kindly asked to signed a consent form. All patients diagnose, age, gender, tooth number were recorded. Patients were then asked to fill four different pain rating scale in an electronic pain rating scale program. Numerical rating scale (NRS) was a scale between "0" and "10", with "0" indicating no pain while "10" indicating worst pain possible. Visual analogue scale (VAS) was a straight line of 10 cm with one end of the line indicated no pain whilst the other end indicated worst pain possible. Color analogue scale (CAS) was the same length of straight line as in VAS with a color change towards to worst pain possible end. Faces rating scale (FRS) consisted of six different faces indicating the level of pain with the first face indicated no pain while the last face indicated worst pain possible. After the patients marked their pain intensity levels in all four scales the results were statistically analyzed to compared the accuracy of four scales with VAS being the golden standard.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic teeth which is in need of root canal treatment

Exclusion Criteria:

* systemic diseases
* age <18 and >80
* being able to understand and accept the study protocol with a written consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
numerical rating scale | through study completion, an average of 1 year
  pain intesity level of patients were recorded on a scale from 0 (no pain) to 10 (worst pain posbile)
visual analogue scale | through study completion, an average of 1 year
  Patients were asked to mark their pain intesity level on a 10 cm line with one end indicating "no pain" and the other end "worst pain possible". The distance between "no pain" and the mark indicates the pain intesity level.
color analogue scale | through study completion, an average of 1 year
  Patients were asked to mark their pain intesity level on a 10 cm color changing line with one end indicating "no pain" and the other end "worst pain possible". The distance between "no pain" and the mark indicates the pain intesity level.
faces rating scale | through study completion, an average of 1 year
  faces rating scale consists of 6 faces with the first face indicating "no pain" and the last face indicating "worst pain possbile"
comparison of four rating scales | through study completion, an average of 1 year
  all four pain rating scales (numerical rating scale, visual analogue scale, color analogue scale, faces rating scale) were compared to analyze correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Tan F EYUBOGLU, PhD, DDS, Study Chair — Assistant Professor
Locations (1):
- Istanbul Medipol University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.

REFERENCES:
- [Result] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- [Result] Price DD, Bush FM, Long S, Harkins SW. A comparison of pain measurement characteristics of mechanical visual analogue and simple numerical rating scales. Pain. 1994 Feb;56(2):217-226. doi: 10.1016/0304-3959(94)90097-3. PMID 8008411
- [Result] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Result] Kremer E, Atkinson HJ, Ignelzi RJ. Measurement of pain: patient preference does not confound pain measurement. Pain. 1981 Apr;10(2):241-248. doi: 10.1016/0304-3959(81)90199-8. PMID 7267140